CLINICAL TRIAL: NCT04406636
Title: Natural History Study in Prodromal and Manifest Huntington Disease Gene Expansion Carriers (HDGECs) - SHIELD HD
Brief Title: Natural History Study in Huntington Disease Gene Expansion Carriers (HDGECs) - SHIELD HD
Acronym: SHIELD HD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TTX N1
Record Dates: First submitted 2020-05-20; First posted 2020-05-28 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Huntington Disease
Keywords: HD
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
SHIELD HD is an international, multisite, prospective, longitudinal cohort natural history study to assess the natural history of HD and its biomarkers that are associated with modulation of the number of cytosine-adenine-guanine (CAG) repeats in the mutant Huntingtin (HTT) gene.

Approximately 60 patients will be enrolled into the study and followed for up to 24 months at clinical sites in North America and Europe.

The results of this study will inform assessments for a future interventional treatment trial.

DETAILED DESCRIPTION:
The rationale for this study is to obtain longitudinal information related to Somatic Instability and DNA damage response genes in HDGECs at various stages of the disease. Established assessments of disease progression will also be recorded.

ELIGIBILITY:
Key Inclusion Criteria

Patients who meet all of the following criteria will be eligible to participate in the study:

1. Capacity to comprehend the study objectives and procedures
2. Documentation of genetically confirmed disease by direct DNA testing, defined as a CAG repeat length ≥39 in the HTT gene
3. Ability to undergo and tolerate MRI scans
4. Ability to tolerate blood draws and lumbar punctures

Key Exclusion Criteria

Patients who meet any of the following criteria will be excluded from participation in the study:

1. Any conditions, including severe chorea and dementia, that would prevent either writing or performing pen and paper, tablet, or computer based tasks as determined by the Investigator
2. Treatment with an investigational drug within 30 days prior to screening or within 5 half lives of the investigational drug, whichever is longer
3. History of gene therapy or cell transplantation or any other experimental brain surgery

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Huntington disease (HD), genetically confirmed by direct DNA testing, either obtained previously or performed at Screening
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
DDR gene expression | 2 years
  To assess deoxyribonucleic acid (DNA) damage repair (DDR) gene expression in accessible biofluids and disease trajectories for established and novel biomarkers and clinical outcomes.

SECONDARY OUTCOMES:
Compare rates of change in biomarkers for disease progression | 2 years
  To compare the rates of change for different outcomes and cytosine adenine guanine (CAG) age product (CAP) Scores.

OTHER OUTCOMES:
Additional biomarkers to be examined | 2 years
  The exploratory objectives of this study are to be determined and may include the examination of additional biomarkers present in CSF, plasma, and whole blood, including but not limited to mutant HTT (mHTT) protein, cytokines, and others, as well as clinical markers of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Rosser, PhD FRCP, Principal Investigator — Cardiff University
Locations (10):
- United States (5):
  - University of California, San Diego (UCSD), San Diego, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Beth Israel Deaconess, Boston, Massachusetts
  - Columbia University, New York, New York
  - Inland Northwest Research, Spokane, Washington
- Canada (2):
  - Centre for Movement Disorders, Toronto, Ontario
  - North York General Hospital, Toronto, Ontario
- ICM - Institut du Cerveau et de la Moelle épinière, Paris, France
- George-Huntington-Institut (GHI), Münster, Germany
- University College London - Institute of Neurology & The National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided